CLINICAL TRIAL: NCT06424405
Title: A New Objective Titration Procedure Using Remotely Intelligent Sleep Monitoring System for the Treatment of Mandibular Advancement Device in OSAHS Patients
Brief Title: A New Objective Titration Procedure for the Treatment of Mandibular Advancement Device in OSAHS Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BeijingJH
Record Dates: First submitted 2024-05-12; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS)
Keywords: Obstructive sleep apnea hypopnea syndrome; Sleep monitoring; contactless sensors; Mandibular advancement device; therapeutic outcomes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- objective titration procedure (Experimental): Objective titration procedure will be based on the objective diagnosis and treatment indicator AHI（Apnea-hypopnea index）which will be provided by RISMS (Remotely intelligent sleep monitoring system). SC-500TM is a comfortable contactless under-mattress sleep monitor, as a main component of the RISMS will be given to patients to collect the sleep data every night at home setting. The sleep report will be generated automatically every day providing the value of AHI and uploaded to the clinicians in real-time. The clinicians will contact the patients by phone every 3-7 days and instruct them remotely to adjust the MAD to increase the mandibular advancement by 0.25-1mm each time, according to AHI together with the self-reported evolution of symptoms. The patients will adapt this new mandibular advancement for 3-7 days and the clinicians will contact them again for further adjustment until a significant improvement of AHI and resolution of symptoms occurs.
  Interventions: Procedure: titration procedure for MAD treatment
- subjective titration procedure (Active Comparator): The subjective titration procedure in this study will be based on self-reported evolution of symptoms and physical limits of the OSAHS patients. Patients will be recalled to the hospital every 1-2 weeks and will be asked about the subjective changes such as snoring, daytime sleepiness，ache of tooth, temporomandibular pain and so on. Then, the clinicians will adjust the MAD to increase degree of mandibular advancement by 0.5-1mm each time. The patients will adapt this new mandibular advancement for 1-2 weeks and have to come back to hospital for further adjustment until an improvement or a resolution of symptoms occurs, or until the patients could not tolerate any further advancement.
  Interventions: Procedure: titration procedure for MAD treatment

INTERVENTIONS:
Procedure: titration procedure for MAD treatment — The OSAHS patients referred for MAD treatment will experience either the objective titration procedure or the subjective titration procedure.

SUMMARY:
The aim of this clinical trial is to apply a new objective titration procedure in obstructive sleep apnea hypopnea syndrome (OSAHS) patients treated with mandibular advancement device (MAD), and to compare this new objective titration procedure with the subjective titration procedure which is commonly used in clinical practice. The remotely intelligent sleep monitoring system (RISMS) will be used in the new objective titration procedure. The main questions it aims to answer are:

1. The efficacy of MAD therapy after each titration procedure.
2. The titration time efficiency and the improvement of subjective symptoms after each titration procedure.

DETAILED DESCRIPTION:
In this study, patients diagnosed with OSAHS and referred for MAD treatment will be recruited. The amount of mandibular protrusion seems to be a key factor in the treatment of MAD. Patients will experience either of the two titration procedures to obtain the optimal mandibular protrusion. One procedure is a new objective titration procedure which will use the RISMS for the treatment of MAD, which will help the clinician instruct the titration according the objective therapeutic indicator. The other procedure is the subjective titration procedure which is commonly used in clinical practice. Finally, the researchers will compare the efficacy of the MAD therapy, the titration time efficiency and the improvement of subjective symptoms between the two titration procedures.

ELIGIBILITY:
Inclusion Criteria:

* OSAHS patients with AHI≥15
* 18≤age≤70 years;
* Subject is capable of giving informed consent
* refusal of or noncompliance with CPAP (continuous positive airway pressure) or unwilling to undergo upper airway surgery
* Normal clinical, periodontal and temporomandibular joint examination

Exclusion Criteria:

* Active periodontal problems including tooth mobility
* active temporomandibular joint dysfunction
* Edentulous patients or Insufficient teeth to support MAD
* patients with severe unstable systemic diseases or suffering from psychiatric disorders
* Enlarged palatine tonsils (Friedman grade IV tonsils)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
efficacy of MAD therapy | The parameter of AHI will be recorded at baseline before the titration and the end of the titration procedures (up to 60 days) using the same PSG device to diagnose OSAHS.
  The efficacy of MAD therapy is in terms of AHI (Apnea-hypopnea index) reduction compared to baseline, as well as the number of responders defined as patients with a reduction in AHI of 50% or more compared to baseline, and/or a follow-up AHI of 10 events/hour or less.

SECONDARY OUTCOMES:
titration time efficiency | The prescribed time is 60 days. The actual titration time is the time taken from the start to the end of the titration procedures (up to 60 days). The saved time is 60 days minus actual titration day.
  The titration time efficiency is the percentage of saved time over the prescribed time.
Epworth sleepiness score(ESS) | ESS will be determined at baseline and the end of titration procedures (up to 60 days).
  The ESS (Epworth Sleepiness Scale) is a self-administered questionnaire that evaluates subjective daytime sleepiness in quotidian situations. The score ranges from 0 to 24 and is usually elevated in sleep apnea patients, indicating a propensity to fall asleep. The score 0 means no sleepiness at daytime, and the score 24 means serious sleepiness. Lower scores mean a better treatment outcome.
Snore Scale(SS） | SS will be determined at baseline and the end of titration procedures (up to 60 days).
  SS （Snore Scale） is measured by A 10-point visual analogue scale (VAS) to assess the severity of snoring, with the VAS ranging from 0, representing no snoring, to 10, causing the bed partner to leave the room or sleep separately. Lower scores mean a better treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Si S Chen, doctor, Study Chair — Beijing Jishuitan Hospital
Locations (1):
- Beijing Jishuitan Hospetal, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No